CLINICAL TRIAL: NCT07404293
Title: Zero CDE Technique for Lens Nucleus Removal During Femtosecond Laser-Assisted Cataract Surgery
Brief Title: Zero CDE Technique for Lens Removal During FLACS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bochner Eye Institute (Other)
Responsible Party: Principal Investigator, Raymond Stein, Medical Director, Bochner Eye Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RS/2024/01 version 2
Record Dates: First submitted 2026-02-05; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Cataract With a Nuclear Sclerosis Grade Between 1 to 3
Keywords: Zero CDE technique; FLACS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cataract removal with Zero CDE technique (Experimental): This is a single-arm, non-comparative, prospective study including cataract patients with a nuclear sclerosis grade between 1 to 3 who desire to undergo cataract surgery and IOL implantation at Bochner Eye Institute, Canada.
  Interventions: Procedure: Femtosecond laser-assisted cataract surgery using Zero CDE

INTERVENTIONS:
Procedure: Femtosecond laser-assisted cataract surgery using Zero CDE — In this single-arm, non-comparative study, patients with cataract grade 1-3 (LOCS III nuclear sclerosis) will undergo cataract removal with the Zero CDE technique that involves no or minimal phaco energy. This is facilitated by a femtosecond laser, which pre-divides the cataractous lens nucleus into multiple small segments that can be aspirated without phaco energy being delivered to the eye.

SUMMARY:
The Zero CDE (cumulative dissipated energy) technique facilitates cataract removal with no or minimal phaco energy. This is facilitated by a femtosecond laser, which pre-divides the cataractous lens nucleus into multiple small segments that can be aspirated without phaco energy being delivered to the eye. In the investigator's experience, this technique consistently shows a stable anterior chamber, a low complication rate, and a rapid return of vision following cataract surgery. This prospective study aims to document the outcomes with the zero CDE technique during femtosecond laser-assisted cataract surgery (FLACS).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over the age of 50 years with operable cataract of nuclear sclerosis grade 1 to 3 as measured by LOCS III grading system (patients with cortical or posterior subcapsular cataract of any grade will be eligible).
* Patients must be able to provide written informed consent for participating in the study.
* Preoperative best corrected visual acuity of 20/25 or worse.

Exclusion Criteria:

* Patients with corneal edema, corneal guttata, pseudoexfoliation, zonular dialysis, or other ocular anomalies (e.g., inflammation, uveitis, previous trauma, suspected microbial infection, glaucoma, and macular disease).
* Patients wearing soft contact lenses will need to discontinue lens wear for 2 weeks, and hard contact lens wearers for one month prior to intraocular lens measurements.
* Women patients of childbearing potential.
* Patients undergoing arcuate keratotomy or other combined surgery with cataract.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2027-03-14 (Estimated); Study Completion 2027-07-14 (Estimated)

PRIMARY OUTCOMES:
% of cataract cases completed with Zero CDE | Intraoperative

SECONDARY OUTCOMES:
Among the cataract cases with zero CDE, o the average amount of balanced salt solution (BSS) (ml) used per case. | Intraoperative
Among the cataract cases with zero CDE o % of cataract cases with corneal edema at one-day postop. | Postoperative Day 1
Among the cataract cases with zero CDE o % of cataract cases with CME at any time up to 3 months postop. | Postoperative 2 weeks, 1 month and 3 months
Among the cases requiring CDE, the amount of phaco energy used | Intraoperative
Incidence of adverse events | Intraoperative, and postoperative Day 1, 2 weeks, 1 month, and 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Bochner Eye Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No